CLINICAL TRIAL: NCT05175053
Title: Early Application of Renal-Replacement Therapy in Patients With Acute Kidney Injury After Cardiac Surgery: A Multicenter Randomized Controlled Trial
Brief Title: Early RRT in AKI After Cardiac Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This multicenter randomized controlled trial planned competitive enrollment across multiple sites; however, no patients were enrolled at one site. Only 44 of 202 participants were enrolled over four years, so early termination is proposed.
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ho Young Hwang, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-2107-213-1239
Record Dates: First submitted 2021-12-10; First posted 2022-01-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Post Cardiac Surgery; Renal Replacement Therapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early RRT group (Experimental): Patients who will undergo renal replacement therapy (RRT) within 6 hours of diagnosis of stage 2 acute kidney injury (AKI).
  Interventions: Other: Renal replacement therapy
- Delayed RRT group (Active Comparator): Patients who will undergo renal replacement therapy (RRT) if one of the absolute indications for RRT is present.
  Interventions: Other: Best medical management

INTERVENTIONS:
Other: Renal replacement therapy — Continuous renal replacement therapy using continuous venovenous hemodiafiltration (CVVHDF)
  Arms: Early RRT group
Other: Best medical management — The best medical management continues until the patient meets absolute indication of renal replacement therapy
  Arms: Delayed RRT group

SUMMARY:
Acute kidney injury (AKI) is one of the major complications after cardiac surgery that may affects 20% to 40% of patients according to the definitions. Also, AKI after cardiac surgery is associated with high morbidity and mortality, with eight-fold increase in the odds ratio of death when renal replacement therapy (RRT) is required. However the indication and the optimal timing of RRT initiation are still controversial.

We hypothesized that a strategy of early initiation of RRT would result in a lower risk of surgical mortality than a standard strategy in post cardiac surgery patients with AKI of Kidney Disease: Improving Global Outcomes (KDIGO) classification stage 2 (serum creatinine, 2.0 times the baseline level; urine output, <0.5mL/kg/h for 6 or more hours).

DETAILED DESCRIPTION:
This trial was designed as a multi-center randomized, controlled trial to recruit 202 patients who develop acute kidney injury (AKI) described as Kidney Disease: Improving Global Outcomes (KDIGO) stage 2 (serum creatinine, 2.0 times the baseline level; urine output, <0.5mL/kg/h for 6 or more hours) after cardiac surgery. Patients were randomized in a 1:1 ratio to 1 of the 2 treatment groups (Early vs. Delayed renal replacement therapy (RRT)) using a computerized system.

Sample size determination : power calculation were performed based on the primary end point (operative mortality). The expected operative mortality in the control group with delayed initiation of RRT was 55% based on the literature. Differences between treatment groups were to be detected with a power of 80%, if the operative mortality of with early initiation of RRT was 35% or less. The expected treatment effect of 20% was calculated on the mortality differences between early and delayed RRT reported in previous studies. A required sample size for the final analysis was 101 patients per treatment group, 202 patients in total (level of significance, α = 0.05; type II error, β= 0.02; potential dropouts= 5%).

Early RRT was initiated within 6 hours of diagnosis of stage 2 AKI.

Delayed RRT was initiated if any one of the following absolute indications for RRT is present

* serum urea level higher than 100mg/dL and/or with uremic encephalopathy
* serum potassium level higher than 6mmol/L and/or with electrocardiography abnormalities
* urine production lower than 0.3mL/kg/hr for 24 hours
* pH of 7.15 or less and/or severe hypotension due to metabolic acidosis
* organ edema in the presence of AKI resistant to diuretic treatment.

The primary end point is operative mortality (described as any death, regardless of cause, occurring (1) within 30 days after surgery in or out of the hospital, and (2) after 30 days during the same hospitalization subsequent to the operation).

The secondary end points included 90 day overall survival, cardiovascular mortality, RRT dependence, and major adverse kidney events (MAKE), adverse events related to RRT or vascular access, duration of mechanical ventilator support and intensive care unit stay, and hospital length of stay.

RRT delivery

: Once RRT was initiated, both groups were treated using continuous venovenous hemodiafiltration (CVVHDF) with identical settings. Initial target dose of hemodiafiltration was 25 to 50mL/kg/hr depends on the decision of attending physician and further adjusted according to the metabolic needs of the patient. Replacement fluid was delivered into the extracorporeal circuit before the filter with a ratio of dialysate to replacement fluid of 1:1. Blood flow was maintained between 100 to 250mL/min. Regional anticoagulation with nafamostat (dosage 20-50mg/hr) was used to prevent circuit clotting if necessary.

RRT was discontinued if renal recovery defined by urine output (>1mL/Kg/hr for 8 hours or more or >1000mL/24h without diuretics; >2000mL/24h with diuretics) and creatinine clearance (>20mL/min) occurred.

If cessation criteria were not fulfilled after 7 days, conversion to intermittent hemodialysis would be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 7 days after cardiac surgery
* Acute kidney injury (AKI) described as Kidney Disease: Improving Global Outcomes (KDIGO) stage 2 (urine output <0.5mL/kg/h for ≥6h or 2-fold increase in serum creatinine compared with baseline)

Exclusion Criteria:

* previous renal replacement therapy
* AKI secondary to obstructive nephropathy
* previous kidney transplantation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2026-02-11 (Actual); Study Completion 2026-02-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with operative mortality | at postoperative 30 days
  any death, regardless of cause, occurring (1) within 30 days after surgery in or out of the hospital, and (2) after 30 days during the same hospitalization subsequent to the operation

SECONDARY OUTCOMES:
Overall survival | at postoperative 90 days
  overall survival
Number of participants with cardiovascular mortality | at postoperative 90 days
  Any death related to cardiac events, including sudden death during follow-up
Number of participants with renal replacement therapy dependency | at postoperative 90 days
  Number of participants who still needs renal replacement therapy at 90 days after operation.
Number of participants with major adverse kidney events (MAKE) | at postoperative 90 days
  MAKE indicates the composite of death, need of renal replacement therapy, and persistent renal dysfunction.
Number of participants with renal replacement therapy related morbidity | at postoperative 90 days
  adverse events related to renal replacement therapy (RRT) or vascular access for RRT.
Duration of mechanical ventilation | at postoperative 30 days
  duration of mechanical ventilator support
Duration of intensive care unit stay | at postoperative 30 days
  duration of intensive care unit stay
Hospital length of stay | at postoperative 30 days
  hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ho Young Hwang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because it is not allowed by our institutional IRB.